CLINICAL TRIAL: NCT01971359
Title: Clinical Outcomes Following Parafascicular Surgical Evacuation of Intracerebral Hemorrhage: A Pilot Study
Acronym: MISPACE
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Andrew Tsung, Andrew Tsung M.D., OSF Healthcare System
Other Study IDs: OSF-13-004
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Intracerebral Hemorrhage
Keywords: Stroke, Intracerebral Hemorrhage, ICH
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hepatitis, Infectious Canine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Retrospective

SUMMARY:
This study is determining the clinical outcomes, based on neurological testing, for the parafascicular minimally invasive clot evacuation technique. We will collect data from the time of surgery up until 90 days post procedure. We will also be looking at financial data as well.

* H(0): there is no economic benefit to the system with early surgical intervention for ICH
* Alternative Hypothesis:H(1) Assuming clinical equipoise, i.e., no benefit in clinical outcome with early surgical intervention (null hypotheses) H(0) is correct), the ability to accelerate the patients care from the entry point to the exit point will result in a significant economic advantage to the system through cost reduction.

DETAILED DESCRIPTION:
Patients will be recruited form the neurology and neurosurgery services at OSF Saint Francis Medical Center. Potential subjects will be identified by the study team which will include all investigators and study coordinators. For those patients who have had the Mi Space procedure, the study team will obtain the patients or patient's surrogate consent for clinical data of hospitalization and follow ups. A secured, de-identified log will be kept of all patients screened, and reasons for exclusion will be documented. Around 65% of unselected patients with ICH (not stratified by baseline predicted risk) have a documented 30 day composite outcome of death or dependency under medical management. Reviews of other types of minimally-invasive ICH surgeries provides data that significantly improved outcomes (meta-analysis odds ratio 0.54(0.39, 0.76)). An odds ratio of 0.54 shows a reduction in risk from 65% to about 50% (15% absolute reduction). Assuming the new procedure is at least as effective than current conventional management, 50 patients provides 66% surety that a 95% 1-sided confidence interval will exclude the chance that the new procedure is worse than medical management. Alternatively, a method of framing this, based on an exact one-sided binomial test of a one-sample proportion and an alpha level of 5%, is that a sample size of 50 patients provides approximately 66% surety/power that the new procedure is superior to medical management (i.e., lower than 65% suffering from death or poor functional outcomes). The critical computed value for this particular test, to provide some initial evidence of superiority, are observing no more than 26 patients (out of 50) suffering from death or dependency under the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria:

* Consecutive patients aged at 18-80 presenting with an acute symptomatic supratertorial primary ICH diagnosed by CT
* Symptom onset to surgery <24 hours (target <8 hours)
* Glascow Coma Score > 9
* Hematoma Volume, between 10ml and 50ml.
* Minimal or no ventricular extension (corresponding to 50% or less of each ventricle)
* NIHSS of >4 or deterioration determined by a neurologist.

Exclusion Criteria:

* Suspected secondary ICH
* Infratentorial ICH
* Isolated IVH
* Uncorrected coagulopathy
* Significant premorbid disability (mRS >1)
* Hydrocephalus
* Contraindication to safe surgical procedure as per neurosurgeon (justification for exclusion on this basis will be recorded)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that present with an ICH at OSF St. Francis Medical Center
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
30-90 day outcomes | 30-90 days
  The primary objective is to compare the 30 day and 90 day clinical outcomes of patients who will undergo parafascicular ICH-evacuation procedure compared to historical outcomes (surgical and non-surgical).

SECONDARY OUTCOMES:
Surgery success rates | 30-90 days
  Another objective will be to describe and quantify peri-operative complications following the parafascicular ICH evacuation. We will assess the success rates of; atraumatic access to the hematoma, effective removal of fibrotic clot by measuring residual hematoma, the ability to achieve hemostasis intra-operatively, and to compare postoperative re-bleeding rates against residual clot volume.

OTHER OUTCOMES:
Financial outcomes | 30-90 days
  We also will be looking at the financial aspect of current medical management and minimally invasive surgeries compared to the parafascicular technique.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tsung, M.D., Principal Investigator — OSF Healthcare System
Locations (1):
- OSF St. Francis Medical Center, Peoria, Illinois, United States